CLINICAL TRIAL: NCT04447573
Title: Immunotherapy With BCMA CAR-T Cells in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Beijing Lu Daopei Hospital (Other); Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCMA CAR-T
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-08

CONDITIONS: Multiple Myeloma
Keywords: BCMA，MM
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CAR-T cells (Experimental): Patients will be treated with BCMA CAR-T cells
  Interventions: Biological: BCMA CAR-T

INTERVENTIONS:
Biological: BCMA CAR-T — Biological: BCMA CAR-T; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis;

SUMMARY:
This study is aimed to evaluate the safety, feasibility and efficacy of BCMA CAR-T in the treatment of relapsed or refractory multiple myeloma

DETAILED DESCRIPTION:
This is a study to evaluate the safety, feasibility and efficacy of BCMA CAR-T in the treatment of relapsed or refractory multiple myeloma.

The Main research objectives:

To evaluate the safety and efficacy of BCMA CAR-T in patients with relapsed or refractory multiple myeloma

The Secondary research objectives:

To investigate the cytokinetic characteristics of BCMA CAR-T in patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study and signed the informed consent form by themselves or their legal guardian;
2. According to the international standard for multiple myeloma (IMWG 2014);
3. Diagnosed as relapsed or refractory multiple myeloma. Relapsed and refractory were defined as follow. Relapsed: patients had received for at least 3 drugs with different mechanisms of action (including protease inhibitors and immunomodulators) and disease progression within 60 days of the most recent treatment. Refractory was defined as: disease progression occurred during the recent treatment, or disease progression occurred within 60 days after treatment;
4. The expression of BCMA in myeloma cells was reported as positive by flow cytometry or immunohistochemistry;
5. No antibody drug was administered within last 2 weeks before cell therapy;
6. ECOG Scores: 0~1
7. Echocardiography showed normal diastolic function, left ventricular ejection fraction (LVEF) ≥ 50%, no serious arrhythmia;
8. The subjects had no pulmonary infection, normal pulmonary function, and indoor air oxygen saturation ≥ 92%;
9. There was no contraindication for peripheral blood sampling;
10. The estimated survival time was more than 12 weeks;
11. The urine pregnancy test of female subjects of childbearing age should be negative and not in lactation; the female or male subjects of childbearing age should take effective contraceptive measures during the whole research process.

Exclusion Criteria:

1. Have a history of allergy to any component of cell products;
2. There are clinically significant cardiovascular diseases, such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or any grade 3 (moderate) or grade 4 (severe) heart disease with cardiac function (according to the functional classification method of the New York Heart AssociationNYHA) with a history of myocardial infarction, angioplasty or stent implantation, unstable angina or other clinically significant heart disease within 12 months before admission;
3. who has suffered from brain injury, consciousness disorder, epilepsy, more serious cerebral ischemia or cerebral hemorrhage disease;
4. Patients who need urgent treatment due to tumor progression or spinal cord compression;
5. The investigator determines that there are serious complications or diseases that will increase the risk of the subject or affect the study, including but not limited to, for example, cirrhosis, recent major trauma, etc;
6. After allogeneic hematopoietic stem cell transplantation;
7. Patients with autoimmune diseases, immunodeficiency or other diseases requiring immunosuppressive （excluding glucocorticoid）therapy;
8. There was uncontrolled active infection;
9. There were live vaccinations within 4 weeks before admission;
10. Active hepatitis (positive for HBVDNA or HCVRNA), syphilis and other acquired and congenital immunodeficiency diseases, including but not limited to those with HIV infection;
11. Subjects had a history of alcohol, drug or mental illness;
12. The researchers believe that there are other conditions that subjects are not suitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after BCMA CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Overall Remission Rate (ORR) | 3 months post CAR-T cells infusion
  Overall Remission Rate (ORR) including partial remission and complete

SECONDARY OUTCOMES:
Efficacy:duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of BCMA CAR- T cells in the genomes of PBMC by qPCR method and percentage of BCMA CAR- T cells measured by flow cytometry method
Cytokine release | First month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&MD, Principal Investigator — Beijing Lu Daopei Hospital
Locations (2):
- China (2):
  - He bei Yan da Lu dao pei Hospital, Yanda, Hebei
  - BeiJing Ludaopei Hospital, Beijing, Yizhuang

REFERENCES:
- [Derived] Zhang XG, Wang L, Yang J, Hu XN, Wang H, Zhang LN, Zhou X, Liu Y, Wang Q, Lu PH. Efficacy and safety of BCMA nanobody CAR T-cell therapy in relapsed or refractory plasma cell myeloma. Blood Adv. 2025 Sep 23;9(18):4543-4552. doi: 10.1182/bloodadvances.2025016322. PMID 40569697